CLINICAL TRIAL: NCT01702194
Title: A Single-Dose, Fixed-Sequence, Two-Period, Two-Treatment Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion of TD-1211 Following an Intravenous Infusion and an Oral Dose of [14C]TD-1211 in Healthy Male Subjects
Brief Title: TD-1211 IV/Oral Mass Balance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0087
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: OIC
Keywords: OIC; Opioid Induced Constipation; Constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Constipation | interventions — Carbon-14; 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-1211 IV [C14] (Experimental): TD-1211 IV [C14]
  Interventions: Drug: TD-1211 IV [C14]
- TD-1211 PO [C14] (Experimental): TD-1211 PO [C14]
  Interventions: Drug: TD-1211 PO [C14]

INTERVENTIONS:
Drug: TD-1211 IV [C14]
  Other Names: TD-1211
  Arms: TD-1211 IV [C14]
Drug: TD-1211 PO [C14]
  Other Names: TD-1211
  Arms: TD-1211 PO [C14]

SUMMARY:
The purpose of this study is to determine TD-1211 is processed by the body.

DETAILED DESCRIPTION:
This study will provide information regarding the metabolic pathway of TD 1211, the need for evaluation of potential drug-drug interactions, the need for studies in special populations and the absolute oral bioavailability of TD-1211. The administration of radiolabeled drug is necessary to fully characterize the rates and routes of elimination of TD 1211, providing further quantitative information on the disposition of TD 1211. The results from this study will allow a more comprehensive comparison between animal and human routes of elimination and metabolic profiles of TD 1211.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, nonsmoking male, 18 to 50 years old, inclusive.
2. Agrees to use a highly effective method of birth control.
3. Body mass index (BMI) 19 to 30 kg/m2, inclusive, and weighs at least 55 kg.
4. Willing and able to give written informed consent.

Exclusion Criteria:

1. Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
2. Hemoglobin <14.1 g/dL or hematocrit < 40.6% at Screening.
3. History of hypersensitivity to drugs, or a history of or any current clinically significant hypersensitivities.
4. Any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas]).
5. Participated in another clinical trial of an investigational drug (or medical device) within 60 days (or 5 half-lives of the investigational drug, whichever is longer) prior to Screening, or is currently participating in another trial of an investigational drug (or medical device).

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | 0 to 168 hours postdose
Peak plasma concentration (Cmax) | 0 to 168 hours postdose
Time to peak plasma concentration (Tmax) | 0 to 168 hours postdose
Half-life (T 1/2) | 0 to 168 hours postdose
Percent total recovery of radioactivity in blood, urine, and feces | 0 to 312 hours postdose

SECONDARY OUTCOMES:
Number of participants with adverse events | Baseline to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Covance, Madison, Wisconsin, United States